CLINICAL TRIAL: NCT01092091
Title: Recombinant Human Arginase I (rhArgI) for Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Study of Pegylated Human Recombinant Arginase for Liver Cancer (BCT-100-002)
Acronym: BCT-100-002
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bio-Cancer Treatment International Limited (Industry)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKCTR-503C; PR/CT0299/2009 (Other: Department of Health, HKSAR)
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Neoplasm; Hepatocellular Carcinoma
Keywords: Neoplasm; Hepatocellular Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — BCT-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-BCT-100 (Experimental): Pegylated Recombinant Human Arginase I
  Interventions: Biological: Pegylated Recombinant Human Arginase I

INTERVENTIONS:
Biological: Pegylated Recombinant Human Arginase I — Weekly dose of PEG-BCT-100 for at least 8 weeks (or until disease progression) at 1600U/kg
  Other Names: PEG-BCT-100

SUMMARY:
The purpose of this study is to determine whether recombinant human arginase (PEG-BCT-100) is safe and effective in the treatment of advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The primary objectives of this study are:

* To evaluate any objective tumor responses to PEG-BCT-100 in HCC patients receiving weekly doses of PEG-BCT-100 alone.
* To perform PK and PD analysis
* To measure Quality of Life of the patients

Secondary objectives of this study are:

* To define any toxicity associated with the metabolic and cellular alterations of ADD relative to dose and PK of PEG-BCT-100 (rhArgIpeg5000).
* To confirm the safety and anti-tumor activity of PEG-BCT-100 at the preferred dose (1600U/kg) in 50 patients (at least 18 evaluable subjects) with advanced HCC.
* To measure duration of response including Overall Survival and Time to Progression analysis

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC according to the European Association for the Study of the Liver criteria
* Known underlying HCC etiology specified by hepatitis B, hepatitis C, post alcoholic cirrhosis, or other
* HCC lesion(s) which are not resectable and which are measurable by C-T scan
* Progression of or non-response of HCC lesions after treatments which are considered best standard of care - surgical resection, radiofrequency ablation, chemoembolization
* No cancer treatment or surgery within the prior 4 weeks, either chemotherapy, targeted biologic or enzymes, either approved or investigational;
* Males or females from 18 to 75 years-old, inclusive;
* Ability and willingness to provide written informed consent;
* Karnofsky performance status of 80% or above and expected survival of more than 12 weeks; and,
* Negative urine pregnancy test, if female, and willingness to use an effective method of contraception during the entire study period
* No cognitive impairment
* Ability to understand and read Chinese

Exclusion Criteria:

* Advancing liver failure indicated by uncontrolled ascites, pleural effusions, encephalopathy, or a Child-Pugh score of C
* Significant hepatic, renal or bone marrow dysfunction indicated by total bilirubin >40 µmol/L, evidence of bile duct obstruction, serum albumin <30 g/L, serum SGOT >5 x upper limit of normal, ANC <1.0 x 10^9/L, platelets <100 x 10^9/L, or INR >2.0
* Significant cardiac or pulmonary disease defined by New York Heart Association (NYHA) Class III or IV, VEF <50% by echo or MUGA, or a history of myocardial infarction within the past 6 months, significant unstable arrhythmia or evidence of ischemia on ECG
* Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Significant active infection including HIV requiring oral or parenteral anti-infective therapies;
* Use of investigational drug(s) within 4 weeks of enrollment; or,
* Prior treatment with arginine depleting agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Tumor response | 12 weeks
  Tumor response endpoints include(a)Objective response for each patient evaluated by RECIST, (b)Modified RECIST criteria will be used as secondary reference, (c) The proportion of patients achieving a partial response or complete response (d) The proportion of patients reporting disease progression by RECIST and the times to progression (e)Serial changes in plasma AFP levels after doses of PEG-BCT-100 and (f)Change in relevant viral serology from baseline to end-of-study

SECONDARY OUTCOMES:
Overall Survival | 12 weeks
  Overall Survival measurement from the date of starting the first dose of PEG-BCT-100 until death from any cause at every 4 weeks until the patient's death, or 3 months from the last patient's study visit, through clinical visits or telephone follow-ups
Time to Progression | 12 weeks
Plasma arginase level | 12 weeks
  The PK endpoints include (a) Dose-related peak to trough concentrations of plasma PEG-BCT-100 over time (b)Plasma clearance of PEG-BCT-100; and(c)Intra- and inter-subject variability of plasma PK parameters to assess the predictability of PEG-BCT-100 administration
Quality of Life | 12 weeks
  Measurement of Quality of Life by completing 2 questionnaires at baseline, week 8 and 4-weekly after week 8 until end of treatment visit. The Chinese version of the EORTC QLQ-C30 will be used, which contains Five functional scales and Three symptom scales. The Chinese version of EORTC QLQ-HCC18 will also be used.
Plasma arginine levels | 12 weeks
  The PD endpoints include (a)The magnitude of plasma arginine depletion relative to the dose (b)The duration of effective ADD assessed by plasma arginine <8 µM relative to the plasma peak and time to clearance (c) The relationships of PEG-BCT-100 dose and its resultant effective ADD to changes in AFP and/or tumor symptoms and measurements(d)The temporal and quantitative relationships of depleted plasma arginine to dose and plasma concentrations of PEG-BCT-100; and (e)Correlation of prolonged arginine depletion with extended survival

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie TP Poon, Prof, Principal Investigator — Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, The University of Hong Kong
Locations (1):
- Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chan SL, Cheng PNM, Liu AM, Chan LL, Li L, Chu CM, Chong CCN, Lau YM, Yeo W, Ng KKC, Yu SCH, Mok TSK, Chan AWH. A phase II clinical study on the efficacy and predictive biomarker of pegylated recombinant arginase on hepatocellular carcinoma. Invest New Drugs. 2021 Oct;39(5):1375-1382. doi: 10.1007/s10637-021-01111-8. Epub 2021 Apr 15. PMID 33856599
- See also: HKCTR-503 — http://www.hkclinicaltrials.com/